CLINICAL TRIAL: NCT07172737
Title: Investigation of the Effects of Functional Inspiratory Muscle Training Applied With Tele-Rehabilitation on Respiratory and Functional Parameters and Quality of Life in Children With Duchenne Muscular Dystrophy: Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Busra Turgut, specialist physiotherapist, Izmir Katip Celebi University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 0451
Record Dates: First submitted 2025-02-04; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: respiratory muscles; tele rehabilitation
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- İntervetion Group 1 (Experimental): IMT will be performed.
  Interventions: Other: Respiratory Muscle Training
- İntervetion group 2 (Experimental): Functional IMT will be performed.
  Interventions: Other: Respiratory Muscle Training
- Control Group (No Intervention): Routine treatment will continue.

INTERVENTIONS:
Other: Respiratory Muscle Training — Respiratory Muscle Training with Telerehabilitation
  Arms: İntervetion Group 1; İntervetion group 2

SUMMARY:
Dushenne muscular dystrophy (DMD), which is characterized by the deficiency of dystrophin protein, prevents the muscle from maintaining its normal activity, causing progressive damage to the heart, respiratory muscles and skeletal muscles. When studies on patients with DMD are examined in the literature, very few studies are found investigating the effectiveness of pure respiratory muscle training, while no studies are found investigating the effectiveness of functional respiratory muscle training.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 5-17
2. Ambulate
3. Having a diagnosis of DMD based on the presence of clinical symptoms, genetic testing or muscle biopsy results
4. Having the ability to perform respiratory function tests
5. Being able to cooperate with the physiotherapist

Exclusion Criteria:

1. Having severe upper extremity contracture or serious systemic disease that would prevent our evaluation
2. Having a respiratory tract infection in the last 3 months
3. Having had an injury or surgery on both upper extremities in the last 6 months

Ages: 5 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Strenght Test | eight week
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurements were used to assess respiratory muscles. MIP and MEP represent the intraoral pressures measured under closed airway conditions during maximal inspiration and expiration, respectively. In this study, these measurements were performed using an intraoral pressure measurement device (Pony FX, COSMED Inc., Rome, Italy) to determine respiratory muscle strength. During the test, for MIP measurement, participants were instructed to perform a maximal inspiration for 1-3 seconds following a maximal expiration while the airway was occluded with a valve. For MEP measurement, after a maximal inspiration, the airway was occluded and participants were asked to perform a maximal expiration for 1-3 seconds. Among the three trials conducted for each parameter, the highest value was recorded.
Respiratory Function Test | eight week
  The measurements were performed using a portable spirometer. In the spirometric assessment, forced expiratory volume in one second (FEV₁), forced vital capacity (FVC), the FEV₁/FVC ratio, and peak expiratory flow (PEF) parameters were examined, and these values were recorded as percentages of the predicted values according to age, height, body weight, and sex.

SECONDARY OUTCOMES:
Modified Medical Research Council (mMRC) Dyspnea Scale | eight weeks
  This scale is a categorical instrument scored from 0 to 4 that assesses the level of breathlessness experienced by patients during daily life activities. Participants responded by selecting one of the five statements that best reflected the severity of their dyspnea.
Six-Minute Walk Test | eight weeks
  The six-minute walk test, frequently used to evaluate physical functional capacity and endurance in neuromuscular diseases, is a submaximal test that measures the walking distance covered by patients over six minutes on a hard surface within a 30-meter corridor. Participants were instructed to walk at their own pace, with rest permitted during the six-minute period, and the total distance walked was recorded in meters.

OTHER OUTCOMES:
Brooke Scale | Baseline
  Upper extremity functions were scored on a scale ranging from 1 (able to abduct arms in a full circle) to 6 (no functional use of the hands).
Vignos Scale | Baseline
  This scale was developed to classify lower extremity functions. Lower extremity functions were scored from 1 (able to walk and climb stairs without assistance) to 10 (confined to bed).

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik training and research hospital, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No